CLINICAL TRIAL: NCT06612580
Title: 68Ga-AAZTA-NI-093 PET/CT: First-in-human Study in Patients With Prostate Cancer
Brief Title: 68Ga-AAZTA-NI-093 PET/CT: First-in-human Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAHFJ-68Ga-AAZTA-NI-093
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PSMA; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-AAZTA-NI-093 PET/ CT (Experimental): 68Ga-AAZTA-NI-093 Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-AAZTA-NI-093. Tracer doses of 68Ga-AAZTA-NI-093 will be used to image lesions of prostate cancer by PET/CT
  Interventions: Drug: 68Ga-AAZTA-NI-093

INTERVENTIONS:
Drug: 68Ga-AAZTA-NI-093 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-AAZTA-NI-093. Tracer doses of 68Ga-AAZTA-NI-093 will be used to image lesions of prostate cancer by PET/CT.

SUMMARY:
68Ga-AAZTA-093 is a novel radiotracer incorporating a hypoxia sensitive nitroimidazole(NI)-moiety and a PSMA-targeting. In this study, we observed the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-AAZTA-NI-093 PET/CT in patients with prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is one of the most common malignancies worldwide in men. Prostate specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. Various low molecular weight radiopharmaceuticals targeting PSMA such as PSMA-11, PSMA-617 for 68Ga- or 177Lu- labeling have been developed. 68Ga-AAZTA-NI-093 is a novel agent incorporating a hypoxia sensitive nitroimidazole(NI)-moiety and a PSMA-targeting. This pilot study was prospectively designed to evaluate the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-AAZTA-NI-093 PET/CT in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated prostate cancer patients;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Within 7 days following PET/CT
  The safety will be assessed by the number and percentage of patients with adverse events; Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry data | through study completion, an average of 3 months
  Calculate the absorbed dose of 68Ga-AAZTA-NI-093 in normal organs.

OTHER OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-AAZTA-NI-093 for prostate cancer in comparison with 68Ga-PSMA-11/68Ga-PSMA-617 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China